CLINICAL TRIAL: NCT02568761
Title: Injection Snoreplasty and Oropharyngeal Exercises: Two Therapeutic Options in the Management of Snoring and Obstructive Sleep Apnea Syndrome.
Brief Title: Injection Snoreplasty and Oropharyngeal Exercises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0637
Record Dates: First submitted 2015-09-15; First posted 2015-10-06 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Snoring; Obstructive Sleep Apnea Syndrome
Keywords: Snoring; Sleep apnea; Obstructive sleep apnea; Speech therapy; Injection snoreplasty; Ethanol; Oropharyngeal exercises
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection snoreplasty (Active Comparator): Nonsurgical treatment involving the injection of 1.5 ml of 50% ethanol (1 ml of 99.5% ethanol diluted in 1ml of 2% xylocaine) into the upper palate. 0.5 ml of the solution will be implemented in three different regions of the submucosal layer of the soft palate, one median and two paramedians.
  Interventions: Procedure: Injection Snoreplasty
- Oropharyngeal Exercises (Active Comparator): Weekly sessions of myofunctional exercises under the supervision of a qualified professional, lasting about 30 minutes each, combined with daily exercises without supervision for a period of three months.
  Interventions: Other: Oropharyngeal Exercises

INTERVENTIONS:
Procedure: Injection Snoreplasty — Nonsurgical treatment involving the injection of 1.5 ml of 50% ethanol (1 ml of 99.5% ethanol diluted in 1ml of 2% xylocaine) into the upper palate.
  Arms: Injection snoreplasty
Other: Oropharyngeal Exercises — Myofunctional isometric and isotonic exercises of the soft palate, pharyngeal side walls, face and tongue.
  Arms: Oropharyngeal Exercises

SUMMARY:
A randomized single blind clinical trial, with a larger sample size than previous studies , to evaluate the effectiveness of injection snoreplasty in the treatment of patients with snoring and obstructive sleep apnea/hypopnea syndrome (OSAHS) compared to oropharyngeal exercises, a low cost therapeutic modality.

DETAILED DESCRIPTION:
34 patients will be randomly allocated into two groups. One group will be submitted to injection snoreplasty and another group will be submitted to daily sessions of oropharyngeal exercises. Researchers involved in interventions will not participate in the outcomes evaluation and researchers responsible for the assessment of outcomes will be blinded to the tested therapeutic modalities.

All patients will be evaluated at a pre-intervention visit, when will be collected objective data and carried out a complete otorhinolaryngological exam. Patients will fill validated specific questionnaires for evaluation of snoring, apnea, daytime sleepiness, fatigue, presence of systemic arterial hypertension and sleep quality. The quality of sleep of the patients bedroom companions will be also evaluated. Patients will be randomized only after these evaluations.

All patients included in the study will be submitted to a portable sleep study. Simultaneously, the objective assessment of snoring will be held, covering the analysis of snoring intensity (measured in decibels) and the snoring index (number of snores per hour of sleep).

Patients allocated to group A will receive injection snoreplasty. Patient returns will be weekly, until the complete healing of the palate. After four weeks of treatment, the bedroom companion will be asked about whether the snoring remains a problem, and if so, the procedure is repeated, with each patient receiving up to three applications. At the end of three months, all evaluations will be repeated and the data obtained will be compared to baseline data.

Patients allocated at group B will be evaluated by a speech therapist. Patients will undergo weekly oropharyngeal exercises sessions under supervision, lasting about 30 minutes each, and will be instructed to perform the exercises daily at home, for a period of three months. At the end of this period, patients will be re-evaluated and the initial data will be compared to the obtained final data.

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated at the Snoring and Apnea Ambulatory of Hospital de Clinicas de Porto Alegre with clinical complaints related to snoring and sleep apnea with polysomnography held within 90 days before the inclusion, evidencing index of apnea/hypopnea from 0 to 30 events per hour of sleep (snoring , mild and moderate apnea), without showing desaturation below 90% for time periods longer than 60 minutes.
* Patient without specific prior treatment for snoring and/or apnea.

Exclusion Criteria:

* Prior pharyngeal surgery to treat snoring or obstructive sleep apnea/hypopnea syndrome (OSAHS).
* Body mass index above 35Kg / m2.
* Nasal or pharyngeal anatomical obstruction higher than 50% of the light.
* Craniofacial deformity.
* Pregnancy.
* Major illnesses associated.
* Ethanol allergy history.
* Absence of a companion to observe the intensity of snoring.
* Patients with no ability to understand the issues (understanding of the proposed procedure and consent form).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Snoring Intensity (measured in decibels) | Three months
Snoring Index (number of snores per hour of sleep) | Three months
Upper airway obstruction | Three months

SECONDARY OUTCOMES:
Sleep quality evaluated with the Pittsburgh Sleep Quality Index | Three months
Sleep quality of the patient room partner evaluated with the Pittsburgh Sleep Quality Index | Three months
Sleepiness (evaluated with the Epworth Sleepiness Scale) | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lavinsky, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Serviço de Otorrinolaringologia do Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel JM. Sleep viewed as a state of adaptive inactivity. Nat Rev Neurosci. 2009 Oct;10(10):747-53. doi: 10.1038/nrn2697. Epub 2009 Aug 5. PMID 19654581
- [Background] Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The Report of an American Academy of Sleep Medicine Task Force. Sleep. 1999 Aug 1;22(5):667-89. No abstract available. PMID 10450601
- [Background] Reimer MA, Flemons WW. Quality of life in sleep disorders. Sleep Med Rev. 2003 Aug;7(4):335-49. doi: 10.1053/smrv.2001.0220. PMID 14505600
- [Background] Drazen JM. Sleep apnea syndrome. N Engl J Med. 2002 Feb 7;346(6):390. doi: 10.1056/NEJM200202073460602. No abstract available. PMID 11832526
- [Background] Chung F, Elsaid H. Screening for obstructive sleep apnea before surgery: why is it important? Curr Opin Anaesthesiol. 2009 Jun;22(3):405-11. doi: 10.1097/ACO.0b013e32832a96e2. PMID 19412094
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Vrints H, Shivalkar B, Hilde H, Vanderveken OM, Hamans E, Van de Heyning P, De Backer W, Verbraecken J. Cardiovascular mechanisms and consequences of obstructive sleep apnoea. Acta Clin Belg. 2013 May-Jun;68(3):169-78. doi: 10.2143/ACB.2981. PMID 24156215
- [Background] Phillipson EA. Sleep apnea--a major public health problem. N Engl J Med. 1993 Apr 29;328(17):1271-3. doi: 10.1056/NEJM199304293281712. No abstract available. PMID 8464440
- [Background] Ellen RL, Marshall SC, Palayew M, Molnar FJ, Wilson KG, Man-Son-Hing M. Systematic review of motor vehicle crash risk in persons with sleep apnea. J Clin Sleep Med. 2006 Apr 15;2(2):193-200. PMID 17557495
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Hoffstein V, Szalai JP. Predictive value of clinical features in diagnosing obstructive sleep apnea. Sleep. 1993 Feb;16(2):118-22. PMID 8446830
- [Background] Zancanella E, Haddad FM, Oliveira LA, Nakasato A, Duarte BB, Soares CF, Cahali MB, Eckeli A, Caramelli B, Drager LF, Ramos BD, Nobrega M, Fagondes SC, Andrada NC; Associacao Brasileira de Otorrinolaringologia e Cirurgia Cervico-Facial; Academia Brasileira de Neurologia; Sociedade Brasileira de Cardiologia; Sociedade Brasileira de Pediatria; Sociedade Brasileira de Pneumologia e Tisiologia. Obstructive sleep apnea and primary snoring: diagnosis. Braz J Otorhinolaryngol. 2014 Jan-Feb;80(1 Suppl 1):S1-16. No abstract available. English, Portuguese. PMID 24838760
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Koskenvuo M, Kaprio J, Telakivi T, Partinen M, Heikkila K, Sarna S. Snoring as a risk factor for ischaemic heart disease and stroke in men. Br Med J (Clin Res Ed). 1987 Jan 3;294(6563):16-9. doi: 10.1136/bmj.294.6563.16. PMID 3101779
- [Background] Schmidt-Nowara WW, Coultas DB, Wiggins C, Skipper BE, Samet JM. Snoring in a Hispanic-American population. Risk factors and association with hypertension and other morbidity. Arch Intern Med. 1990 Mar;150(3):597-601. doi: 10.1001/archinte.150.3.597. PMID 2310278
- [Background] Norton PG, Dunn EV. Snoring as a risk factor for disease: an epidemiological survey. Br Med J (Clin Res Ed). 1985 Sep 7;291(6496):630-2. doi: 10.1136/bmj.291.6496.630. PMID 3928056
- [Background] Hoffstein V. Blood pressure, snoring, obesity, and nocturnal hypoxaemia. Lancet. 1994 Sep 3;344(8923):643-5. doi: 10.1016/s0140-6736(94)92084-2. PMID 7915347
- [Background] Yeboah J, Redline S, Johnson C, Tracy R, Ouyang P, Blumenthal RS, Burke GL, Herrington DM. Association between sleep apnea, snoring, incident cardiovascular events and all-cause mortality in an adult population: MESA. Atherosclerosis. 2011 Dec;219(2):963-8. doi: 10.1016/j.atherosclerosis.2011.08.021. Epub 2011 Aug 22. PMID 22078131
- [Background] Marshall NS, Wong KK, Cullen SR, Knuiman MW, Grunstein RR. Snoring is not associated with all-cause mortality, incident cardiovascular disease, or stroke in the Busselton Health Study. Sleep. 2012 Sep 1;35(9):1235-40. doi: 10.5665/sleep.2076. PMID 22942501
- [Background] Lee SA, Amis TC, Byth K, Larcos G, Kairaitis K, Robinson TD, Wheatley JR. Heavy snoring as a cause of carotid artery atherosclerosis. Sleep. 2008 Sep;31(9):1207-13. PMID 18788645
- [Background] Beninati W, Harris CD, Herold DL, Shepard JW Jr. The effect of snoring and obstructive sleep apnea on the sleep quality of bed partners. Mayo Clin Proc. 1999 Oct;74(10):955-8. doi: 10.4065/74.10.955. PMID 10918859
- [Background] Collop NA. Portable monitoring for the diagnosis of obstructive sleep apnea. Curr Opin Pulm Med. 2008 Nov;14(6):525-9. doi: 10.1097/MCP.0b013e328312ed4a. PMID 18812829
- [Background] Brietzke SE, Mair EA. Injection snoreplasty: how to treat snoring without all the pain and expense. Otolaryngol Head Neck Surg. 2001 May;124(5):503-10. doi: 10.1067/mhn.2001.115400. PMID 11337652
- [Background] Schwab RJ, Pasirstein M, Pierson R, Mackley A, Hachadoorian R, Arens R, Maislin G, Pack AI. Identification of upper airway anatomic risk factors for obstructive sleep apnea with volumetric magnetic resonance imaging. Am J Respir Crit Care Med. 2003 Sep 1;168(5):522-30. doi: 10.1164/rccm.200208-866OC. Epub 2003 May 13. PMID 12746251
- [Background] Sher AE, Schechtman KB, Piccirillo JF. The efficacy of surgical modifications of the upper airway in adults with obstructive sleep apnea syndrome. Sleep. 1996 Feb;19(2):156-77. doi: 10.1093/sleep/19.2.156. PMID 8855039
- [Background] Nordgard S, Stene BK, Skjostad KW. Soft palate implants for the treatment of mild to moderate obstructive sleep apnea. Otolaryngol Head Neck Surg. 2006 Apr;134(4):565-70. doi: 10.1016/j.otohns.2005.11.034. PMID 16564373
- [Background] Friedman M, Schalch P, Lin HC, Kakodkar KA, Joseph NJ, Mazloom N. Palatal implants for the treatment of snoring and obstructive sleep apnea/hypopnea syndrome. Otolaryngol Head Neck Surg. 2008 Feb;138(2):209-16. doi: 10.1016/j.otohns.2007.10.026. PMID 18241718
- [Background] Powell NB, Riley RW, Troell RJ, Li K, Blumen MB, Guilleminault C. Radiofrequency volumetric tissue reduction of the palate in subjects with sleep-disordered breathing. Chest. 1998 May;113(5):1163-74. doi: 10.1378/chest.113.5.1163. PMID 9596289
- [Background] Gunawardena I, Robinson S, MacKay S, Woods CM, Choo J, Esterman A, Carney AS. Submucosal lingualplasty for adult obstructive sleep apnea. Otolaryngol Head Neck Surg. 2013 Jan;148(1):157-65. doi: 10.1177/0194599812461750. Epub 2012 Sep 26. PMID 23014996
- [Background] Guimaraes KC, Drager LF, Genta PR, Marcondes BF, Lorenzi-Filho G. Effects of oropharyngeal exercises on patients with moderate obstructive sleep apnea syndrome. Am J Respir Crit Care Med. 2009 May 15;179(10):962-6. doi: 10.1164/rccm.200806-981OC. Epub 2009 Feb 20. PMID 19234106
- [Background] STRAUSS JF. A new approach to the treatment of snoring: A preliminary report. Arch Otolaryngol.1943 Sep;38(3):225-9.
- [Background] Brietzke SE, Mair EA. Injection snoreplasty: extended follow-up and new objective data. Otolaryngol Head Neck Surg. 2003 May;128(5):605-15. doi: 10.1016/S0194-59980300229-8. PMID 12748553
- [Background] Iseri M, Balcioglu O. Radiofrequency versus injection snoreplasty in simple snoring. Otolaryngol Head Neck Surg. 2005 Aug;133(2):224-8. doi: 10.1016/j.otohns.2005.04.018. PMID 16087019
- [Background] Al-Jassim AH, Lesser TH. Single dose injection snoreplasty: investigation or treatment? J Laryngol Otol. 2008 Nov;122(11):1190-3. doi: 10.1017/S0022215108002648. Epub 2008 Jun 9. PMID 18538040
- [Background] Lorenzetti FTM. Injeção roncoplástica: comparação entre etanol 50% e oleato de etanolamina 5% no tratamento do ronco [Internet] [text]. Universidade de São Paulo; 2011. At http://www.teses.usp.br/teses/disponiveis/5/5143/tde-20072011-151743/
- [Background] Labra A, Haro-Valencia R, Huerta-Delgado AD, Jimenez-Correa U, Sanchez-Narvaez F. Efficacy of submucosal sodium tetradecyl sulfate in the soft palate as a treatment of the mild obstructive sleep apnea syndrome: a pilot study. Sleep Disord. 2012;2012:597684. doi: 10.1155/2012/597684. Epub 2012 Jan 24. PMID 23471094
- [Background] Puhan MA, Suarez A, Lo Cascio C, Zahn A, Heitz M, Braendli O. Didgeridoo playing as alternative treatment for obstructive sleep apnoea syndrome: randomised controlled trial. BMJ. 2006 Feb 4;332(7536):266-70. doi: 10.1136/bmj.38705.470590.55. Epub 2005 Dec 23. PMID 16377643
- [Background] Guimarães KCC. Efeitos dos exercícios orofaríngeos em pacientes com apnéia obstrutiva do sono moderada: estudo controlado e randomizado [Internet] [text]. Universidade de São Paulo; 2008. At: http://www.teses.usp.br/teses/disponiveis/5/5150/tde-22082008-170703/
- [Background] Friedman M, Ibrahim H, Joseph NJ. Staging of obstructive sleep apnea/hypopnea syndrome: a guide to appropriate treatment. Laryngoscope. 2004 Mar;114(3):454-9. doi: 10.1097/00005537-200403000-00013. PMID 15091218